CLINICAL TRIAL: NCT00934388
Title: A Randomised, Blinded Study on Laparoscopic Mesh Reinforcement for Chronic Groin Pain.
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Royal Hobart Hospital (Other Government)
Responsible Party: Mr. Stuart Walker, Royal Hobart Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SRW 001
Record Dates: First submitted 2009-07-07; First posted 2009-07-08 (Estimated); Last update posted 2010-03-16 (Estimated); Status verified 2010-03

CONDITIONS: Chronic Groin Pain
Keywords: Sportsmans groin, Gilmores groin
MeSH Terms: interventions — Laparoscopy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mesh placed in pre peritoneal plane (Experimental)
  Interventions: Procedure: Pre peritoneal mesh placement
- No mesh placed (Active Comparator)
  Interventions: Procedure: Laparoscopy

INTERVENTIONS:
Procedure: Pre peritoneal mesh placement
  Arms: Mesh placed in pre peritoneal plane
Procedure: Laparoscopy
  Arms: No mesh placed

SUMMARY:
Chronic groin pain is a frequent cause for referral to general surgeons. In some cases this pain may be due to the presence of a hernia. However, if on clinical examination there is no palpable lump or bulge, the cause of the pain may be difficult to elucidate. Some of these patients may have the diagnosis of sportsman's groin. Other names which have been attached to this condition include Gilmores groin and sportsmans hernia. These conditions are more commonly associated with sportsmen and women but those who do not play sport may also receive this diagnosis. Sportsman's groin is thought to be a syndrome of weakness of the posterior inguinal wall without a clinically recognisable hernia. Differing explanations for sportsman's groin include avulsion of the conjoint tendon from the pubic tubercle, weakening of the transversalis fascia, tears in the internal or external oblique, superficial inguinal ring dilatation and abnormalities of the rectus abdominus insertion.

There is some evidence that pre peritoneal mesh placement in these patients may be beneficial. The theory being that the mesh prevents pressure transmission to the damages structures, allowing them to heal more rapidly.

Aim. To assess the potential benefit of pre peritoneal mesh placement using the TAPP technique in patients with chronic groin pain.

ELIGIBILITY:
Inclusion Criteria:

* Groin pain (unilateral or bilateral) for at least 4 months. In this way, patients with temporary symptoms will be excluded from undergoing unnecessary surgery.
* Tenderness over pubic tubercle or superficial inguinal ring.

Exclusion Criteria:

* Aged less than 18 years Aged more than 50 years - due to increased incidence of sacro-iliac and hip pathology.
* Bulge, lump or cough impulse consistent with inguinal or femoral hernia on clinical examination.
* Patients unwilling or unable to provide informed consent. Medically unfit for general anaesthetic
* Pregnant women
* Diabetes - due to diabetic neuropathy
* Steroid use
* QST suggestive of nerve entrapment.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2011-01; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Return to normal activities | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Hobart Hospital, Hobart, Tasmania, Australia